CLINICAL TRIAL: NCT01060579
Title: A Phase 2, Double-masked, Randomized, Active-controlled, Dose-response Study Assessing the Safety and Ocular Hypotensive Efficacy of AR-12286 in Patients With Elevated Intraocular Pressure
Brief Title: Study of AR-12286 Versus Latanoprost in Patients With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR-12286-CS202
Record Dates: First submitted 2010-01-30; First posted 2010-02-02 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-04

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — AR-12286; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AR-12286 0.5% ophthalmic solution (Experimental)
  Interventions: Drug: AR-12286 0.5% ophthalmic solution
- AR-12286 0.25% Ophthalmic Solution (Experimental)
  Interventions: Drug: AR-12286 0.25% Ophthalmic solution
- Latanoprost 0.005% ophthalmic solution (Experimental)
  Interventions: Drug: Latanoprost ophthalmic solution

INTERVENTIONS:
Drug: AR-12286 0.5% ophthalmic solution — q.d. PM
  Arms: AR-12286 0.5% ophthalmic solution
Drug: AR-12286 0.25% Ophthalmic solution — q.d. PM
  Arms: AR-12286 0.25% Ophthalmic Solution
Drug: Latanoprost ophthalmic solution — q.d. PM
  Other Names: Xalatan(R)
  Arms: Latanoprost 0.005% ophthalmic solution

SUMMARY:
A 28 day study of the safety and efficacy of two concentrations of topical AR-12286 in treating ocular hypertension and open-angle glaucoma compared to latanoprost. Hypothesis: The ocular hypotensive efficacy of each dose of AR-12286 ophthalmic solution will not be different from that of an active control.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT) and currently being treated with ocular hypotensive medication.
3. Unmedicated (post-washout) IOP ≥ 22 mm Hg at 2 eligibility visits (07:00-09:00 hr), 2-7 days apart.
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
5. Has used a commercially available IOP-lowering medication in one or both eyes for at least 30 days over the 90 days prior to the screening visit.
6. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic (in either eye):

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure. Note: Previous laser peripheral iridotomy is acceptable.
2. Intraocular pressure > 36 mm Hg
3. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s).
5. Refractive surgery in study eye(s) (e.g., radial keratotomy, PRK, LASIK, etc.).
6. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months.
7. History or evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at baseline (Visit 1), or of herpes simplex keratitis
8. Contact lens wear within 30 minutes of instillation of study medication.
9. Ocular medication of any kind within 30 days of Visit 1, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 1) or c) lubricating drops for dry eye (which may be used throughout the study).
10. Clinically significant ocular disease (e.g. corneal edema, uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (i.e., cup-disc ratio > 0.8).
11. Central corneal thickness greater than 600 μ.
12. Any abnormality preventing reliable applanation tonometry of either eye.

Systemic:

1. Clinically significant abnormalities in laboratory tests at screening.
2. Clinically significant systemic disease (e.g., uncontrolled diabetes, myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
3. Participation in any investigational study within the past 30 days.
4. Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
5. Due to status of preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the mean intraocular pressure (IOP) across subjects within treatment group on each day at each post-treatment timepoint | 28 days of dosing

SECONDARY OUTCOMES:
Mean change from diurnally adjusted baseline IOP at each timepoint | 28 days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Thomas van Haarlem, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (18):
- United States (18):
  - United Medical Research Institute, Inglewood, California
  - North Bay Eye Associates, Petaluma, California
  - Centre For Health Care, Poway, California
  - East Florida Eye Institute, Stuart, Florida
  - Marvin Greenberg, MD, Tamarac, Florida
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Bradley Kwapiszeski, MD, Shawnee Mission, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Comprehensive Eye Care, St Louis, Missouri
  - Mount Sinai School Of Medicine, New York, New York
  - Rochester Ophthalmology Group, Rochester, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Charlotte Eye Ear Nose and Throat, Charlotte, North Carolina
  - The Eye Institute, Tulsa, Oklahoma
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Univ Eye Surgeons, Maryville Ctr., Maryville, Tennessee
  - Texan Eye, Austin, Texas
  - Medical Center Ophth. Associates, San Antonio, Texas